CLINICAL TRIAL: NCT07063121
Title: Evaluation of a Digital Application and a Guide for Promoting Subjective Well-Being and Resilience in Colombian Youths: A Randomized Clinical Trial
Brief Title: App-Based Intervention for Youth Well-Being and Resilience in Colombia
Acronym: ShEdge-COL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Centro Internacional de Educación y Desarrollo Humano (Other)
Collaborators: The Digging Deep Project (Unknown); Fondation Botnar (Switzerland) (Unknown)
Responsible Party: Principal Investigator, Sara Victoria Alvarado Salgado, General Director of CINDE, Fundación Centro Internacional de Educación y Desarrollo Humano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SE-GSEA
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Promotion; Subjective Well-Being; Emotional Resilience
Keywords: Digital mental health; Mobile health intervention; Subjective well-being; Emotional resilience; Youth mental health; Behavioral intervention; App-based intervention

STUDY DESIGN:
Intervention Model Description: This study used a three-arm parallel assignment design to evaluate the effects of a digital mental health intervention. Participants were randomized into one of three groups: (1) Shadow's Edge app only, (2) Shadow's Edge app plus a printed Guide to Self-Awareness (GSEA), and (3) a waitlist control group. The interventions were delivered concurrently across groups over an 8-week period. The control group did not receive the intervention during the initial data collection phase but was given access to both the app and the guide after their second assessment. No crossover occurred during the intervention period. All participants completed repeated measures at regular intervals. This model allowed for the evaluation of short-term changes in subjective well-being and resilience, and the comparison of intervention effects between groups. Random assignment was conducted using computerized allocation and stratified to ensure balance in sex and age distribution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App only (Experimental): Participants in this arm used only the Shadow's Edge mobile application. They were instructed to engage with the app for at least 20 minutes per day over an 8-week period. The app promotes emotional expression, self-reflection, and resilience through a narrative-based experience that includes writing prompts and creative activities.
  Interventions: Behavioral: Shadow's Edge mobile app
- App + Guide (Experimental): Participants in this arm used both the Shadow's Edge mobile application and the printed Guide to Self-Awareness (GSEA). The intervention was delivered over 8 weeks, with daily use of the app and weekly completion of guided reflection activities. The guide was designed to enhance emotional insight, mindfulness, and social-emotional skills.
  Interventions: Behavioral: Shadow's Edge mobile app; Behavioral: Guide to Self-Awareness (GSEA)
- Waitlist Control (No Intervention): Participants in this arm did not receive the intervention during the first two assessments. They were evaluated at two timepoints without access to the app or guide. After the second assessment, they received access to both the Shadow's Edge app and the GSEA for ethical and comparative purposes.

INTERVENTIONS:
Behavioral: Shadow's Edge mobile app — A mobile application adapted for Colombian youth that uses interactive storytelling, journaling, and emotional regulation activities to promote subjective well-being and resilience.
  Arms: App + Guide; App only
Behavioral: Guide to Self-Awareness (GSEA) — A printed guide developed to promote emotional insight, mindfulness, self-awareness, and social-emotional skills through structured reflection activities. Designed to be used alongside the Shadow's Edge app.
  Arms: App + Guide

SUMMARY:
This study evaluated the effectiveness of a mobile application called Shadow's Edge, with or without a printed self-awareness guide, in improving well-being and emotional resilience among Colombian youth aged 18 to 22. A total of 184 participants were randomly assigned to three groups: one used the app only, another used both the app and the guide, and a control group received delayed access. Participants completed psychological assessments before and after the intervention. The main outcomes included changes in well-being and resilience measured with standardized scales. Results showed that the app improved well-being and resilience in the short term. However, adding the guide did not produce additional benefits. The study highlights the potential of digital mental health tools in promoting emotional well-being among young people in low- and middle-income countries.

DETAILED DESCRIPTION:
This study is a randomized clinical trial designed to evaluate the effectiveness of a mobile mental health application (Shadow's Edge) and a printed self-awareness guide (GSEA - Guide to Self-Awareness) in improving subjective well-being and emotional resilience among Colombian youth. The study was conducted in response to the growing demand for accessible, evidence-based mental health tools in low- and middle-income countries (LMICs), where structural barriers such as inequality, poverty, and conflict limit access to traditional mental health services. The COVID-19 pandemic further highlighted the need for remote, scalable solutions to address emotional well-being in youth populations.

Shadow's Edge is a narrative-based digital tool developed by the nonprofit Digging Deep Project. It combines principles from narrative therapy, positive psychology, and existential psychology. Through writing prompts and creative expression in a post-apocalyptic fictional setting, users are guided to explore their emotions and build resilience. The game environment fosters engagement by allowing users to rebuild a city devastated by a storm-a metaphor for personal adversity. It has been previously evaluated in different contexts, with promising results in mental health promotion and resilience-building among adolescents.

The Guide to Self-Awareness (GSEA), developed as a printed complement to the app, incorporates socio-emotional learning strategies to deepen reflection. It includes structured exercises that promote mindfulness, emotional regulation, goal-setting, empathy, and communication skills. Both tools were culturally adapted to the Colombian context between 2021 and 2022, involving feedback from local adolescents and youth leaders.

A total of 305 young people expressed interest in the study through an open call disseminated via youth organizations. From these, 210 met the eligibility criteria and were randomized into three groups using the randomizeR package in R. The eligibility criteria included being between 18 and 22 years old, residing in Colombia for at least 6 months, and not being regular users of high-action video games (based on guidance from the app developers, who indicated that such users may have lower engagement with narrative-based tools). Participants with prior experience using Shadow's Edge were excluded. The final sample included 184 participants.

The groups were structured as follows:

App Group: Participants used Shadow's Edge only.

App + Guide Group: Participants used Shadow's Edge and completed exercises from the GSEA.

Control Group (Waitlist): Participants received delayed access to both tools after a second baseline measurement.

Data were collected using three validated instruments:

* WHO-5 Well-Being Index (Campo-Arias et al., 2015 - Colombian validation): Measures subjective well-being over the last two weeks using five items on a Likert scale.
* Abbreviated Resilience Scale (EAR) (Rodríguez-Rey et al., 2016 - Spanish validation): A six-item scale assessing perceived resilience.
* Abbreviated Resilient Coping Scale (EAAR) (Trejos-Herrera et al., 2023 - Colombian validation): A four-item scale measuring resilient coping behaviors.

Measurements were taken in person at baseline and at 4 and 8 weeks for the intervention groups. The control group was evaluated four times: twice prior to gaining access to the tools and twice after. All instruments were administered in print. Compliance with the app usage was monitored via daily digital progress logs and backend usage data linked to anonymous codes. Participants were encouraged to use the app for at least 20 minutes daily.

Statistical analysis was conducted using mixed-effects regression models in R, controlling for group assignment, age, sex, and the number of words written in the app journal (used as a proxy for engagement). The analysis aimed to determine changes over time in each outcome measure, as well as between-group differences.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 22 years at the time of enrollment
* Resided in Colombia for at least 6 months prior to the start of the study
* Provided informed consent to participate
* Not a frequent user of high-action video games (e.g., first-person shooter or battle royale formats)
* Had not previously used the Shadow's Edge mobile application

Exclusion Criteria:

* Any participant sharing a household or close familial relationship with another enrolled participant (to prevent contamination across study arms)
* Failure to meet any of the inclusion criteria

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Change in WHO-5 Well-Being Index Score | Baseline (Week 0), Week 4, and Week 8
  The WHO-5 Well-Being Index is a 5-item self-report scale developed by the World Health Organization to assess subjective psychological well-being over the past two weeks. Each item is rated on a 6-point Likert scale ranging from 0 ("At no time") to 5 ("All of the time"). Total scores range from 0 to 25, with higher scores indicating better well-being. The instrument has been validated in Colombia (Campo-Arias et al., 2015) and is widely used in clinical trials. Changes in scores across the three measurement points (baseline, 4 weeks, and 8 weeks) will be used to assess the effectiveness of the intervention.

SECONDARY OUTCOMES:
Change in Abbreviated Resilience Scale (EAR) Score | Baseline (Week 0), Week 4, and Week 8
  The Abbreviated Resilience Scale (EAR) is a 6-item self-report measure used to assess perceived resilience, including the ability to recover from stress. Each item is rated on a 5-point Likert scale. Total scores range from 6 to 30, with higher scores indicating greater resilience. The Spanish version validated in Colombia (Rodríguez-Rey et al., 2016) was used in this study. Scores were collected at baseline, week 4, and week 8 to assess changes in resilience across time and study groups.
Change in Abbreviated Resilient Coping Scale (EAAR) Score | Baseline (Week 0), Week 4, and Week 8
  The Abbreviated Resilient Coping Scale (EAAR) is a 4-item self-report measure designed to assess resilient coping behavior under stress. Each item is rated on a 5-point Likert scale, yielding total scores ranging from 4 to 20. Higher scores indicate stronger coping ability. The Colombian validation by Trejos-Herrera et al. (2023) was used in this study. Scores were obtained at three time points to analyze improvements in coping strategies over time.

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Scoppetta, Ph.D., Study Director — Fundación Centro Internacional de Educación y Desarrollo Humano
Locations (1):
- Sede Bogotá, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes (WHO-5, EAR, and EAAR scores), collected at all time points.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available beginning 6 months after publication of the main findings and for up to 5 years thereafter.
Access Criteria: Data will be made available to qualified researchers upon reasonable request for purposes consistent with the original study objectives. A data use agreement will be required.